CLINICAL TRIAL: NCT04021953
Title: Evaluation of eHealth Videos for the Singaporean Gay, Bisexual and Queer Male Community
Brief Title: The People Like Us Evaluation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: National Centre for Infectious Diseases, Singapore (Unknown); Action for AIDS Singapore (Unknown)
Responsible Party: Principal Investigator, TAN KAY JIN RAYNER, Principal Investigator, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S-19-059
Record Dates: First submitted 2019-07-12; First posted 2019-07-16 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: HIV/AIDS; Sexually Transmitted Infection; Homosexuality; Health Behavior; Stigma, Social; Health Care Seeking Behavior
Keywords: HIV Testing; STI Testing; Homophobia; eHealth; Singapore
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases; Homosexuality; Health Behavior; Social Stigma; Patient Acceptance of Health Care; Homophobia | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The online intervention comprises a series of six videos, each about 10-minutes in length, entitled the People Like Us series. The intervention was developed by gayhealth.sg and Action for AIDS Singapore in 2018. The series follow the love and sex lives of four ethnically-diverse GBQ men of varying socioeconomic backgrounds, as they negotiate issues of sexual health, mental health, and relationships throughout the six-part miniseries.
  The intervention group will also be provided with an e-pamphlet on sexual wellness catered to GBMSM. This e-pamphlet has been developed by the National Skin Centre and Department of Sexually Transmitted Infections Clinic specifically for information on sexual wellness among GBMSM. It comprises segments on HIV/STI symptoms, etiology, information on how to seek help for HIV/STI, behavioral and biomedical methods of HIV prevention.
  Interventions: Behavioral: People Like Us Online Video Series Intervention; Behavioral: Sexual Health Pamphlet (Standard of Care)
- Control Group (Active Comparator): The control group will be provided with an e-pamphlet on sexual wellness catered to GBMSM. This e-pamphlet has been developed by the National Skin Centre and Department of Sexually Transmitted Infections Clinic specifically for information on sexual wellness among GBMSM. It comprises segments on HIV/STI symptoms, etiology, information on how to seek help for HIV/STI, behavioral and biomedical methods of HIV prevention.
  Interventions: Behavioral: Sexual Health Pamphlet (Standard of Care)

INTERVENTIONS:
Behavioral: People Like Us Online Video Series Intervention — People Like Us miniseries incorporates key sexual health messages to:
  1. Increase viewers' knowledge and perceptions of HIV and other STI risk;
  2. Address homophobia and sexual orientation disclosure;
  3. Increase safer-sex negotiation self-efficacy;
  4. Promote positive attitudes towards condom use and other safe sex behaviors;
  5. Build skills and self-efficacy for practicing safer sex;
  6. Provide information on HIV and other STI testing and its benefits;
  7. Provide information on resources for HIV/STI testing and other mental health services;
  8. Model appropriate behaviors around practicing safer sex.
  Each video in the six-part series ends with an educational video segment featuring the managers of Action for AIDS and Gayhealth.sg, who provide a brief synopsis of the episode and cover key points relevant to mental and sexual health for GBQ men.
  Arms: Intervention Group
Behavioral: Sexual Health Pamphlet (Standard of Care) — The control group will be provided with an e-pamphlet on sexual wellness catered to GBMSM. This e-pamphlet has been developed by the National Skin Centre and Department of Sexually Transmitted Infections Clinic specifically for information on sexual wellness among GBMSM. It comprises segments on HIV/STI symptoms, etiology, information on how to seek help for HIV/STI, behavioral and biomedical methods of HIV prevention.

SUMMARY:
The study is a pragmatic, randomized controlled trial design to evaluate an online video series developed by a community-based organization in Singapore for gay, bisexual and queer men.

A total of 300 HIV-negative, gay, bisexual and queer men in Singapore aged 18 to 29 years old will be recruited with the assistance of the partner community-based organization (CBO), Action for AIDS Singapore. Recruitment will utilize both online and offline channels, and with the help of other CBOs in Singapore. Participants should also not have watched the video prior to their participation in this study, which will be ascertained through a questionnaire.

Participants will subsequently be randomized into the intervention arm (n=150) and the control arm (n=150). The treatment group (n=150) will be assigned the intervention along with sexual health information via a pamphlet, while the control group (n=150) will be assigned only the sexual health information via a pamphlet. This will be conducted through block randomization.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported HIV-negative status, or unsure of HIV status
* Self-reported gay, bisexual or queer sexual orientation
* Self-reported male gender, regardless of sex assigned at birth
* Self-reported age of 18 to 29 years old at point of recruitment
* Singapore citizen or permanent resident at the point of recruitment
* Self-reported as never having watched an online video drama series by Gayhealth.sg or Action for AIDS in the last year

Exclusion Criteria:

* Participants who have watched the People Like Us Series prior to study
* Participants who have self-reported being HIV-positive
* Participants who are not English-literate
* Participants aged below 18 or above 29 at baseline recruitment

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Self-identified Male gender (regardless of sex assigned at birth)
Enrollment: 300 (Actual)
Dates: Start 2019-10-13 (Actual); Primary Completion 2020-07-06 (Actual); Study Completion 2020-07-06 (Actual)

PRIMARY OUTCOMES:
Change in intention to test for HIV at 3 months | 3 months
  Participants are asked: "How likely are you to get tested for HIV in the next three months?"; to which they may respond:
  1. Extremely unlikely to get tested
  2. Very unlikely to get tested
  3. Somewhat unlikely to get tested
  4. Somewhat likely to get tested
  5. Very likely to get tested
  6. Extremely likely to get tested
Change in intention to test for HIV at 6 months | 6 months
  Participants are asked: "How likely are you to get tested for HIV in the next three months?"; to which they may respond:
  1. Extremely unlikely to get tested
  2. Very unlikely to get tested
  3. Somewhat unlikely to get tested
  4. Somewhat likely to get tested
  5. Very likely to get tested
  6. Extremely likely to get tested
Change in intention to test for Syphilis at 3 months | 3 months
  Participants are asked: "How likely are you to get tested for Syphilis in the next three months?"; to which they may respond:
  1. Extremely unlikely to get tested
  2. Very unlikely to get tested
  3. Somewhat unlikely to get tested
  4. Somewhat likely to get tested
  5. Very likely to get tested
  6. Extremely likely to get tested
Change in intention to test for Syphilis at 6 months | 6 months
  Participants are asked: "How likely are you to get tested for Syphilis in the next three months?"; to which they may respond:
  1. Extremely unlikely to get tested
  2. Very unlikely to get tested
  3. Somewhat unlikely to get tested
  4. Somewhat likely to get tested
  5. Very likely to get tested
  6. Extremely likely to get tested
Change in intention to test for Chlamydia and Gonorrhea at 3 months | 3 months
  Participants are asked: "How likely are you to get tested for Chlamydia and Gonorrhea in the next three months?"; to which they may respond:
  1. Extremely unlikely to get tested
  2. Very unlikely to get tested
  3. Somewhat unlikely to get tested
  4. Somewhat likely to get tested
  5. Very likely to get tested
  6. Extremely likely to get tested
Change in intention to test for Chlamydia and Gonorrhea at 6 months | 6 months
  Participants are asked: "How likely are you to get tested for Chlamydia and Gonorrhea in the next three months?"; to which they may respond:
  1. Extremely unlikely to get tested
  2. Very unlikely to get tested
  3. Somewhat unlikely to get tested
  4. Somewhat likely to get tested
  5. Very likely to get tested
  6. Extremely likely to get tested
HIV testing at 3 months | 3 months
  Participants are asked: "When did you go for you last (most recent) voluntary HIV test?"; to which they may respond:
  1. Never
  2. In the last 3 months
  3. In the last 6 months
  4. 6 to 12 months ago
  5. More than 1 year ago
HIV testing at 6 months | 6 months
  Participants are asked: "When did you go for you last (most recent) voluntary HIV test?"; to which they may respond:
  1. Never
  2. In the last 3 months
  3. In the last 6 months
  4. 6 to 12 months ago
  5. More than 1 year ago
Syphilis testing at 3 months | 3 months
  Participants are asked: "When did you go for you last (most recent) voluntary Syphilis test?"; to which they may respond:
  1. Never
  2. In the last 3 months
  3. In the last 6 months
  4. 6 to 12 months ago
  5. More than 1 year ago
Syphilis testing at 6 months | 6 months
  Participants are asked: "When did you go for you last (most recent) voluntary Syphilis test?"; to which they may respond:
  1. Never
  2. In the last 3 months
  3. In the last 6 months
  4. 6 to 12 months ago
  5. More than 1 year ago
Chlamydia and Gonorrhea testing at 3 months | 3 months
  Participants are asked: "When did you go for you last (most recent) voluntary Chlamydia or Gonorrhea test?"; to which they may respond:
  1. Never
  2. In the last 3 months
  3. In the last 6 months
  4. 6 to 12 months ago
  5. More than 1 year ago
Chlamydia and Gonorrhea testing at 6 months | 6 months
  Participants are asked: "When did you go for you last (most recent) voluntary Chlamydia or Gonorrhea test?"; to which they may respond:
  1. Never
  2. In the last 3 months
  3. In the last 6 months
  4. 6 to 12 months ago
  5. More than 1 year ago
Self-reported regularity of HIV testing at 3 months | 3 months
  Participants are asked: "On average, how regularly do you test for HIV?"; to which they may respond:
  1. I do not test regularly
  2. Once every few years
  3. Once a year
  4. Once every 6 months
  5. Once every 3 months
  6. Once a month
Self-reported regularity of HIV testing at 6 months | 6 months
  Participants are asked: "On average, how regularly do you test for HIV?"; to which they may respond:
  1. I do not test regularly
  2. Once every few years
  3. Once a year
  4. Once every 6 months
  5. Once every 3 months
  6. Once a month
Self-reported regularity of Syphilis testing at 3 months | 3 months
  Participants are asked: "On average, how regularly do you test for Syphilis?"; to which they may respond:
  1. I do not test regularly
  2. Once every few years
  3. Once a year
  4. Once every 6 months
  5. Once every 3 months
  6. Once a month
Self-reported regularity of Syphilis testing at 6 months | 6 months
  Participants are asked: "On average, how regularly do you test for Syphilis?"; to which they may respond:
  1. I do not test regularly
  2. Once every few years
  3. Once a year
  4. Once every 6 months
  5. Once every 3 months
  6. Once a month
Self-reported regularity of Chlamydia and Gonorrhea testing at 3 months | 3 months
  Participants are asked: "On average, how regularly do you test for Chlamydia and Gonorrhea?"; to which they may respond:
  1. I do not test regularly
  2. Once every few years
  3. Once a year
  4. Once every 6 months
  5. Once every 3 months
  6. Once a month
Self-reported regularity of Chlamydia and Gonorrhea testing at 6 months | 6 months
  Participants are asked: "On average, how regularly do you test for Chlamydia and Gonorrhea?"; to which they may respond:
  1. I do not test regularly
  2. Once every few years
  3. Once a year
  4. Once every 6 months
  5. Once every 3 months
  6. Once a month

SECONDARY OUTCOMES:
Risk perception for HIV | 3 months and 6 months
  Risk perception is measures through a questions (slider scale) that asks participants: "How much risk do you think you are at of getting HIV?". Participants will rate this from 0 to 10 (0=no risk at all; 10=very high risk)
Risk perception for other sexually transmitted infections | 3 months and 6 months
  Risk perception is measures through a questions (slider scale) that asks participants: "How much risk do you think you are at of getting other sexually transmitted infections?". Participants will rate this from 0 to 10 (0=no risk at all; 10=very high risk)
Knowledge of HIV Pre-Exposure Prophylaxis | 3 months and 6 months
  Participants are tested on their knowledge of HIV Pre-Exposure Prophylaxis by providing a response (1=True; 2=False; 3=I do not know) to two questions:
  "HIV Pre-Exposure Prophylaxis is an effective means of preventing HIV infection". The correct answer is "True".
  "HIV Pre-Exposure Prophylaxis can also reduce the chances of acquiring other STIs". The correct answer is "False".
  Each correct answer provides a score of 1 point.
Knowledge of risks associated with acquiring other sexually transmitted infections | 3 months and 6 months
  Participants are tested on their knowledge of other sexually transmitted infections by providing a response (1=True; 2=False; 3=I do not know) to three questions:
  "Gonorrhea can be transmitted through oral sex". The correct answer is "True".
  "Chemsex, or the use of substances during sex, often increases a person's risk of engaging in risky sexual behavior and acquiring HIV or other STIs" The correct answer is "True".
  "There is a/are clinics in Singapore where I can test anonymously for HIV and Syphilis". The correct answer is "True".
  Each correct answer provides a score of 1 point.
Knowledge of HIV | 3 months and 6 months
  Participants are tested on their knowledge of HIV by providing a response (1=True; 2=False; 3=I do not know) to two questions:
  "An HIV-positive individual who has achieved viral suppression or an 'undetectable' viral load has almost zero chances of transmitting the virus to someone else through sexual intercourse". The correct answer is "True".
  "An HIV-positive individual on effective treatment can live a long, healthy, and productive life". The correct answer is "True".
  Each correct answer provides a score of 1 point.
Connectedness to LGBT Community | 3 months and 6 months
  This is an 8-item scale adapted from Frost & Meyer (2012) that measures a participant's self-perceived connectedness to the LGBT community on a 4-point Likert Scale. The measure is a sum score of all 8 items.
Modified Self-Concealment Scale | 3 months and 6 months
  This is a 7-item scale adapted from Scrimshaw (2013) that measures a participant's self-concealment of their sexual orientation on a 5-point Likert Scale. The measure is a sum score of all 7 items.
Consistent condom use for anal sex with casual partners or sex workers | 3 months and 6 months
  This is assessed by the question, "In the last 3 months, how often did you use a condom when having anal sex with a casual partner?" or "In the last 3 months, how often did you use a condom when having anal sex with a sex worker/money boy?" (Options are always, more than half the time, about half the time, less than half the time, never used a condom). Participants who give the answer 'Always' are classified as having consistent condom usage for anal sex with causal partners or sex workers.
Incidence of sexually transmitted infections | 3 months and 6 months
  This is defined as self-reporting a diagnosis of Syphilis, Chlamydia, Genital Herpes, Genital Warts, Hepatitis C, or Gonorrhea at the 3-month or 6-month follow-up.
Perceived Homophobia | 3 months and 6 months
  This is a 6-item scale adapted from Smolenski, Ross, Risser, and Rosser (2009) that measures a participant's self-concealment of their sexual orientation. The measure is a sum score of all 6 items.
Internalized Homophobia | 3 months and 6 months
  This is a 5-item scale adapted from Frost and Meyer (2013) that measures a participant's internalized homophobia on a 4-point Likert Scale. The measure is a sum score of all 5 items.
HIV testing self-efficacy | 3 months and 6 months
  This is a 10-item scale adapted from Jamil and colleagues (2015) that measures a participant's self-efficacy in HIV testing on a 5-point Likert Scale. The measure is a sum score of all 10 items.
HIV testing social norms | 3 months and 6 months
  This is a 9-item scale adapted from Pettifor and colleagues (2010) that measures a participant's perceptions on norms around HIV testing on a 4-point Likert Scale. The measure is a sum score of all 9 items.

CONTACTS AND LOCATIONS:
Overall Officials: Rayner Kay Jin Tan, B.Soc.Sci, Principal Investigator — National University of Singapore
Locations (1):
- National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tan RKJ, Koh WL, Le D, Banerjee S, Chio MT, Chan RKW, Wong CM, Tai BC, Wong ML, Cook AR, Chen MI, Wong CS. Effect of a Popular Web Drama Video Series on HIV and Other Sexually Transmitted Infection Testing Among Gay, Bisexual, and Other Men Who Have Sex With Men in Singapore: Community-Based, Pragmatic, Randomized Controlled Trial. J Med Internet Res. 2022 May 6;24(5):e31401. doi: 10.2196/31401. PMID 35522470
- [Derived] Tan RKJ, Koh WL, Le D, Tan A, Tyler A, Tan C, Banerjee S, Wong CS, Wong ML, Chio MT, Chen MI. Effect of a web drama video series on HIV and other sexually transmitted infection testing among gay, bisexual and queer men: study protocol for a community-based, pragmatic randomised controlled trial in Singapore: the People Like Us (PLU) Evaluation Study. BMJ Open. 2020 Apr 7;10(4):e033855. doi: 10.1136/bmjopen-2019-033855. PMID 32269026